CLINICAL TRIAL: NCT06973122
Title: Effect of Combined Paragastric Autonomic Neural Blockade and Laparoscopic Assisted Transversus Abdominis Plane Block on Visceral Pain After Bariatric Surgery
Brief Title: Paragastric Neural Blockade and Laparoscopic Assisted Transversus Abdominis Plane Block on Visceral Pain After Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, sarah mohamed, lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 0307254
Record Dates: First submitted 2025-05-06; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Visceral Pain
Keywords: paragastric; bariatric surgery; visceral pain
MeSH Terms: conditions — Visceral Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paragastric and transversus abdominis plane block (Experimental): patients will undergo laparoscopic bariatric surgery under general anesthesia, paragastric autonomic neural blockade and laparoscopic assisted transversus abdominis plane block
  Interventions: Procedure: combined paragastric autonomic neural blockade and laparoscopic assisted transversus abdominis plane block
- Transversus abdominis plane block (Other): patients will undergo laparoscopic bariatric surgery under general anesthesia and laparoscopic assisted transversus abdominis plane block
  Interventions: Procedure: laparoscopic assisted transversus abdominis plane block

INTERVENTIONS:
Procedure: combined paragastric autonomic neural blockade and laparoscopic assisted transversus abdominis plane block — paragastric autonomic neural blockade and laparoscopic assisted transversus abdominis plane block
  Other Names: group C
  Arms: Paragastric and transversus abdominis plane block
Procedure: laparoscopic assisted transversus abdominis plane block — laparoscopic assisted transversus abdominis plane block
  Other Names: group P
  Arms: Transversus abdominis plane block

SUMMARY:
after laparoscopic bariatric surgery, visceral pain (VP) remains a significant issue. VP causes autonomic symptoms, such as nausea and vomiting, and does not respond to conventional pain management methods that target incisional pain. The present study was performed to test the effect of use of combined paragastric autonomic neural blockade and laparoscopic assisted transversus abdominis plane block on visceral pain during laparoscopic bariatric surgery and in the early postoperative period.

DETAILED DESCRIPTION:
Visceral pain (VP) is the main cause of pain in the first 24 hours after laparoscopic bariatric surgery (LBS) and other laparoscopic surgeries, although being rarely acknowledged.(1) Traditional pain management regimens do not effectively address patients' visceral, colicky pain following LBS. Patients often describe VP as epigastric and retrosternal pain. This occurs immediately after LBS, peaks at 24 hours, and can extend up to 72 hours.(2) More than 65% of patients with VP after LBS experience autonomic symptoms, including nausea, retching, and vomiting. These symptoms are the leading cause of readmission within 30 days.(3, 4)

The management of postoperative visceral pain is challenging and frequently necessitates the use of opioids. Additionally, postoperative nausea and vomiting (PONV) continues to be the primary cause of prolonged hospital stays and readmissions.(5) Visceral sensory pathways are dispersed both centrally and peripherally. The stomach is mostly dependent on external neural inputs, especially parasympathetic and sympathetic pathways, although having intrinsic neural plexuses that grant it considerable autonomy. Afferent pathways of the sympathetic nervous system are located at the celiac ganglion, and they mostly have an inhibitory effect on the muscles and motility of the stomach. On the other hand, the vagus nerve and its branches, which make up the parasympathetic nervous system, primarily have an excitatory effect on the tone and motility of the stomach.(6)

Autonomic nerve blocks have been discussed in pain management literature. In particular, celiac ganglion blocks have been utilized to treat chronic pain brought on by pancreatitis or foregut cancers. Neuraxial blocks have been shown to be a secure and successful way to treat chronic pain in these patients. Nevertheless, as far as we know, No perioperative multimodal pain treatment algorithms have included paragastric autonomic neural blockade (PG-ANB) in gastrointestinal surgery. It is suggested that this autonomic blockade works primarily through two mechanisms: a decrease in the parasympathetic control over the stomach, whereby reverses the elevated muscle tone, deactivates the organ wall's mechanosensitive receptors, and blocks the afferent sympathetic fibers that send VP to the spinal cord.(7,8)

There is a paucity in studies about use of PG-ANB in pain control after bariatric surgery. Our hypothesis is that use of paragastric autonomic neural blockade in laparoscopic bariatric surgery may relieve postoperative visceral pain and decrease the incidence of postoperative nausea and vomiting.

Aim of the work:

The present study aims to test the effect of use of combined paragastric autonomic neural blockade and laparoscopic assisted transversus abdominis plane block on visceral pain during laparoscopic bariatric surgery and in the early postoperative period.

Primary outcome:

• Postoperative pain score

Secondary outcomes:

* Intraoperative fentanyl requirements
* Postoperative nalbuphine requirements
* Time to first dose of rescue analgesia
* Postoperative nausea and vomiting

Patients :

Study settings:

This study will be conducted in general surgery department, Alexandria university hospitals.

Study design:

Double blind, randomized, prospective and controlled study

Sample size calculation:

The sample size was calculated using G*Power software based on a preliminary study. Assuming a medium effect size (Cohen's d = 0.5) to detect a clinically meaningful difference between the two groups, a power of 80%, and a significance level of 0.05 (two-tailed), a total of 120 participants (60 in each group) were required.

Parameter Value Description Study Design Two-group comparison Para gastric autonomic nerve blockade with TAP block vs. TAP block only.

Statistical Test Independent t-test Assuming continuous outcome data. Effect Size (Cohen's d) 0.5 Medium effect size (assumed in the absence of pilot data).

Power (1 - β) 80% Probability of detecting a true effect if it exists. Alpha (α) 0.05 Significance level (two-tailed). Allocation Ratio 1:1 Equal sample sizes in both groups. Sample Size per Group 60 Number of participants required in each group. Total Sample Size 120 Total number of participants required for the study.

Study population:

All patients will be randomized 1:1 using a sealed envelope method. Patients will be divided into two equal groups:

Group C: patients will undergo laparoscopic bariatric surgery under general anesthesia, paragastric autonomic neural blockade and laparoscopic assisted transversus abdominis plane block

Group T: patients will undergo laparoscopic bariatric surgery under general anesthesia and laparoscopic assisted transversus abdominis plane block

Inclusion criteria:

1. Age: 20-50 years, both sexes.
2. ASA physical status class I to III.
3. BMI 35- 50 kg/m²

Exclusion criteria:

1. Severe cardiac disorder
2. chronic renal failure
3. liver cirrhosis
4. allergy to bupivacaine
5. patients with history of chronic opioid consumption
6. HBA1C > 7%

Methods:

Preoperative evaluation and preparation:

During preoperative visit, evaluation of patients will be carried out through proper history taking, clinical examination and routine laboratory investigations including complete blood picture, coagulation profile, blood urea, serum creatinine, serum electrolytes, fasting blood glucose, glycosylated haemoglobin (HBA1C), liver function tests and any other investigation needed.

Pre-anesthetic preparation and premedication:

* Informed written consent, from all individual participants who will be included in this study will be taken during preoperative visit.
* Patients should be trained during preoperative visit on a visual analogue scale (VAS), with 0 corresponding to no pain and 10 to the worst pain imaginable.
* Patients will be informed about the analgesic regimen
* Thrombotic prophylaxis (enoxaparin 40 mg) will be started 12 hours before surgery.

On arrival to operative theatre, intravenous cannula will be inserted and standard monitoring will be established using multichannel monitor (Carescape Monitor B650, GE Healthcare Finland) to monitor the following in both groups:

* Electrocardiogram (ECG) for heart rate and rhythm. (Beats/min).
* Non-invasive measurement of arterial blood pressure. (Mean blood pressure in mmHg).
* Pulse oxygen saturation. (SpO2%).
* End tidal CO2 tension (in mmHg).
* Entropy

Anesthesia:

After preoxygenation for 3 minutes, anesthesia will be induced in both groups with propofol 2mg/kg of lean body weight until loss of verbal response, fentanyl 2µg/kg and atracurium 0.5 mg/kg intravenously. Anesthesia will be maintained by isoflurane with 50% oxygen in air (1.2-1.5 %) to maintain entropy between 40-60. Mechanical ventilation will be performed with tidal volume of 8 ml/ kg and a respiratory rate of 12-15 cycles/min to maintain the end-tidal carbon dioxide tension between 35 and 40 mmHg and an oxygen saturation of ≥ 98 per cent with 50 percent oxygen in air. Incremental doses of atracurium will be given every 30 minutes to maintain muscle relaxation. In both groups, signs of insufficient analgesia (eg, tachycardia over 20% of the preoperative value occur during anesthesia) or somatic response (eg, movement ,tearing ,or sweating), will be treated with additional boluses of fentanyl 0.5 mcg/kg intraoperatively as needed. Intraoperatively, all patients will receive IV dexamethasone (8 mg), paracetamol (1 g), ketorolac (30 mg).

After induction of general anesthesia , patients in group T will receive laparoscopically assisted bilateral transversus abdominis plane block, while patients in group c will receive paragastric autonomic neural blockade in addition to laparoscopic assisted transversus abdominis plane block.

Technique of laparoscopic transversus abdominis plane block:(9) For each side, 20 ml of 0.25 % bupivacaine will be injected in the middle of iliac crest and costal margin in midaxillary line . 14-gauge needle will be inserted from the skin until sudden decrease in resistance will be felt, corresponding to the external oblique fascia. To ensure that the needle will not go beyond the peritoneum, laparoscopy will be used to observe the formation of a bulge at the back of the transversus abdominis muscle.

Technique of paragastric autonomic neural blockade:(10) The paragastric lesser omentum neural block will be performed with a 25-gauge short needle attached to a venous catheter extension introduced through the left 12-mm port. The needle will be capped during its introduction, and the cap will be removed inside the abdomen using a grasper and kept under direct vision at all times. Infiltration of 20 mL of thick 0.5% bupivacaine will be performed at six levels in the fatty tissue of the paragastric area with careful aspiration preceding the infiltration of fluid. Proper infiltration of the lesser omentum along the vagus nerve and distal branches at the esophagogastric junction, proximal stomach, mid-stomach, and distal antrum should be ensured. Next, the area overlying the hepatic artery will be infiltrated. Finally, the area overlying the left gastric artery will be infiltrated in the posterosuperior paragastric area by elevating the proximal half of the sleeve from the stomach's neo-greater curvature. The cap will be then reapplied to the needle, and the assembly will be removed from the abdominal cavity.

At the end of surgery, awake extubation, in a semi-sitting position, will be done. Then, the patient will be transferred to the PACU. In PACU, all patients will be assessed for presence and severity of pain; using Visual Analog Scale (VAS). Patients will be prescribed IV nalbuphine 0.15 mg/kg of lean body weight boluses on 4-6 hours basis with a maximum of 20 mg if VAS > 3. Pain control in the ward will be achieved with IV paracetamol 1 g every 6 hours and ketorolac 30 mg every 12 hours. Outcome assessors in PACU and ward will be blinded to patient group assignment and to the nature of the study.

Measurements:

The following data will be measured:

I- Demographic data:

Patient's age (years), sex, body mass index (BMI) (kg/m2 ) and co-morbidities will be recorded.

II- Haemodynamic measurements:

* Pulse rate (Beat / min).
* Non-invasive measurement of mean arterial blood pressure (in mmHg) All previous parameters will be continuously monitored and recorded before induction of anesthesia, prior to performance of the block , 10 minutes after performance of block and at 1, 12 h in the postoperative period III- Assessment of pain using VAS at 4, 8, 12 and 24 hours postoperatively. IV- Number of patients who need opioids at 4, 8 and 12 h in the postoperative period V- Postoperative nausea and vomiting VI- time to first dose of rescue analgesia VII- Intraoperative staple line bleeding

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-50 years, both sexes.
* ASA physical status class I to III.
* BMI 35- 50 kg/m²

Exclusion Criteria:

* Severe cardiac disorder
* chronic renal failure
* liver cirrhosis
* allergy to bupivacaine
* patients with history of chronic opioid consumption
* HBA1C > 7%

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-04-04 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
postoperative pain score | postoperative day 1
  VAS score

SECONDARY OUTCOMES:
Number of patients who need opioids in postoperative period | postoperative day 1
  number
time to first dose of rescue analgesia | postoperative day1
  minutes
Postoperative nausea and vomiting | postoperative day 1
  number

CONTACTS AND LOCATIONS:
Overall Officials: sarah m elgamal, MD, Principal Investigator — Alexandria University
Locations (1):
- Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Daes J, Morrell DJ, Hanssen A, Caballero M, Luque E, Pantoja R, Luquetta J, Pauli EM. Paragastric Autonomic Neural Blockade to Prevent Early Visceral Pain and Associated Symptoms After Laparoscopic Sleeve Gastrectomy: a Randomized Clinical Trial. Obes Surg. 2022 Nov;32(11):3551-3560. doi: 10.1007/s11695-022-06257-9. Epub 2022 Sep 2. PMID 36050617